CLINICAL TRIAL: NCT06255834
Title: A Phase 1, Randomized, Double-blind, Placebo-controlled, Single and Multiple Dose Escalation Study to Evaluate the Safety, Tolerability, Pharmacokinetics (PK) and Food Effect of Orally Administered IPG11406 in Healthy Adult Participants
Brief Title: Phase 1 Study for IPG11406 in Health Volunteer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Nanjing Immunophage Biotech Co., Ltd (Industry)
Collaborators: Zhejiang Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: IPG11406-C001
Record Dates: First submitted 2023-12-25; First posted 2024-02-13 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Inflammatory Bowel Diseases
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double (Participant, Investigator)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (9):
- Cohort 1 (SAD - 0.5 mg) (Experimental): 4 subjects in this cohort will receive a single dose of IPG11406 0.5 mg qd and 2 subjects will receive a single dose of placebo 0.5 mg qd orally.
  Interventions: Drug: IPG11406
- Cohort 2 (SAD - 2 mg) (Experimental): 4 subjects in this cohort will receive a single dose of IPG11406 2 mg qd and 2 subjects will receive a single dose of placebo 2 mg qd orally.
  Interventions: Drug: IPG11406
- Cohort 3 (SAD - 6 mg) (Experimental): 4 subjects in this cohort will receive a single dose of IPG11406 6 mg qd and 2 subjects will receive a single dose of placebo 6 mg qd orally.
  Interventions: Drug: IPG11406
- Cohort 4 (SAD - 20 mg) (Experimental): 6 subjects in this cohort will receive a single dose of IPG11406 20 mg qd and 2 subjects will receive a single dose of placebo 20 mg qd orally.
  Interventions: Drug: IPG11406
- Cohort 5 (SAD - 40 mg) (Experimental): 6 subjects in this cohort will receive a single dose of IPG11406 40 mg qd and 2 subjects will receive a single dose of placebo 40 mg qd orally.
  Interventions: Drug: IPG11406
- Cohort 6 (SAD - 80 mg) (Experimental): 6 subjects in this cohort will receive a single dose of IPG11406 80 mg qd and 2 subjects will receive a single dose of placebo 80 mg qd orally.
  Interventions: Drug: IPG11406
- Cohort 7 (MAD - 10 mg) (Experimental): 6 subjects in this cohort will receive a dose of IPG11406 10 mg qd and 2 subjects will receive a dose of placebo 10 mg qd orally from Day 1 to 10-day.
  Interventions: Drug: IPG11406
- Cohort 8 (MAD - 20 mg) (Experimental): 6 subjects in this cohort will receive a dose of IPG11406 20 mg qd and 2 subjects will receive a dose of placebo 20 mg qd orally from Day 1 to 10-day.
  Interventions: Drug: IPG11406
- Cohort 9 (MAD - 40 mg) (Experimental): 6 subjects in this cohort will receive a dose of IPG11406 40 mg qd and 2 subjects will receive a dose of placebo 40 mg qd orally from Day 1 to 10-day.
  Interventions: Drug: IPG11406

INTERVENTIONS:
Drug: IPG11406 — IPG11406 Activity: An antagonist of the GPR183 Dosage form: Tablet Strength: 0.5 mg, 10 mg and 40 mg Storage：15 ~ 25 °C in a tightly sealed container, protect from light Administration: In each cohort, IPG11406 or placebo tablets are orally administered once on Day 1 (Part A) or daily for 10 days from Day 1 to Day 10 (Part B) in a fasted state. Oral doses will be administered with 240 ml of water. Tablets should not be chewed or crushed.
  Participants in the FE Cohort will receive a second single dose of IPG11406 following a standardized high fat meal upon ≥4 days washout period after the first dose.
  IPG11406 Placebo Placebo tablets: tablets identical to IPG11406 tablets
  Other Names: IPG11406 Placebo

SUMMARY:
A phase 1, randomized, double-blind, placebo-controlled, single and multiple dose escalation study to evaluate the safety, tolerability, pharmacokinetics (PK) and food effect of orally administered IPG11406 in healthy adult participants

DETAILED DESCRIPTION:
This is a phase 1, randomized, double-blind, placebo-controlled, single and multiple dose escalation study to evaluate the safety, tolerability, PK and food effect of orally administered IPG11406 in healthy adult participants. The study will involve two sequential parts: a single ascending dose (SAD) period (Part A) followed by a multiple ascending dose (MAD) period (Part B).

Part A Dose escalation will start from 0.5 mg. Currently, the 6 dose cohorts are Cohort 1 (0.5 mg), Cohort 2 (2 mg), Cohort 3 (6 mg), Cohort 4 (20 mg), Cohort 5 (40 mg), Cohort 6 (80 mg). About 42 healthy adult participants are being sequentially enrolled in 6 cohorts.

There are 6 participants in Cohort 1 to Cohort 3. In each cohort, 4 participants will receive IPG11406 and 2 participants will receive the placebo as per the randomization code.

Approximately 8 participants will be enrolled in Cohort 4 to Cohort 6 respectively; in each cohort, 6 participants will receive IPG11406 and 2 participants will receive the placebo as per the randomization code.

In each Cohort, 2 sentinel participants will be dosed at least 48 hours prior to the remaining participants. One sentinel will be dosed with IPG11406 and the other with a matching placebo. The remaining participants will be dosed only if no significant safety issues are identified in the sentinel participants. Doses and sampling intervals may be modified based on the PK and safety data that emerges throughout the study.

One of the SAD (Cohort 5 is tentatively to be selected, it may be modified based on the decision of SMC meeting.) cohorts will be selected to assess the effect of food on the pharmacokinetic parameters and referred to as the food effect (FE) cohort. Participants in this cohort will be requested to return to the clinical site to receive a second dose of IPG11406 or placebo after the administration of a meal, upon completion of the 4-day safety follow up period after their first dose. The second dose of IPG11406 or placebo will be administered following a standardized high fat meal (total calories approximately 800 to 1000 calories, with approximately 50% of total calories from fat).

Healthy participants will be screened within 28 days prior to dosing. Participants in the SAD cohorts (including FE cohort) will be admitted to the study site on Day -1 for a total of 6 days. Administration of a single dose of IPG11406 or the placebo will occur on Day 1 under fasted conditions (Following an overnight fast of at least 10 hours, subjects will receive a single dose of IPG11406 or placebo with 240 mL water. Water can be ingested as desired except for 1 hour pre-dose until one hour post dose.). Participants will be discharged on Day 5 following collection of samples for PK analyses and the completion of safety assessments. A follow-up visit will occur on Day 8.

Participants in the FE cohort will be admitted to the study site for at least 10 days for the 2 administrations of IPG11406. A washout of ≥ 4 days will be included between investigational product (IP) administrations. Administration of a single dose of IPG11406 or placebo will occur on Day 1 under fasted condition, and Day 6 (anticipated) under postprandial condition. Following completion of all safety assessments and sampling for PK analyses, subjects will be discharged on Day 10 (anticipated) after the second dose. There will be a follow-up visit on Day 13 (anticipated) after the single dose administration in each period.

Once the final participant in the cohort has completed the Day 5 assessments and been discharged, the Safety Monitoring Committee (SMC) will review cumulative blinded safety data (including follow-up visit data from preceding cohorts) and available PK data to determine the safety and tolerability of the study drug. If the dose level is determined to be safe and well-tolerated, the next dose cohort will be enrolled and randomized in preparation to receive the next dose level of IPG11406 or the placebo.

Part B Three dose levels (10 mg, 20 mg and 40 mg) are anticipated to be evaluated in the MAD, once daily. There will be approximately 8 subjects per cohort, 6 subjects will receive IPG11406 and 2 subjects will receive placebo per the randomization code.

For Cohort M1 (10 mg), the MAD phase will commence following the establishment of the safety and tolerability of Cohort 4 (20 mg) in the SAD. The SMC will evaluate the safety, tolerability and PK data obtained from the participants of cohort 4 in the SAD to determine if the Cohort M1 will be enrolled and randomized to receive the 10 mg multiple dose levels of IPG11406 or placebo.

For Cohort M2 (20 mg), the SMC will evaluate the safety, tolerability and PK data obtained from the participants of cohort 5 (40 mg) in the SAD as well as the safety and PK data from Cohort M1 to determine if the Cohort M2 will be enrolled and randomized to receive the 20 mg multiple dose levels of IPG11406 or placebo.

For Cohort M3 (40 mg), the SMC will evaluate the safety, tolerability and PK data obtained from the participants of cohort 6 (80 mg) in the SAD as well as the safety and PK data from Cohort M2 to determine if the Cohort M3 will be enrolled and randomized to receive the 40 mg multiple dose levels of IPG11406 or placebo.

All subjects will be screened within 28 days prior to dosing and will be admitted to the study site on Day -1. Dosing will start on the morning of Day 1 and will continue over a 10-day period at each dose level. Blood draws will be collected for the assessment of PK parameters. Participants will be discharged on Day 14 following completion of all PK sample collection and safety assessments. There will be a follow-up visit 7 days after the last dose.

Once the final participant in the cohort has completed the Day 14 assessments and been discharged, the SMC will review blinded cumulative safety data (including the follow-up visit data) and available PK data to determine the safety and tolerability of the study drug.

ELIGIBILITY:
Inclusion Criteria:

Participants must meet all of the following criteria to be included in the study:

Demography

1. Healthy adult male or female participants between 18 and 55 years of age (inclusive).
2. Body weight between 45 and 100 kg (inclusive) and body mass index (BMI) within 18~32 kg/m2 (inclusive).

   Health status
3. In good health as determined by screening tests. Good health is defined as having no clinically relevant abnormalities identified by a detailed medical history, full physical examination (including measurement of blood pressure and pulse rate), 12-lead ECG, and clinical laboratory tests.

   * Vital signs ( measured after resting for 5 minutes semi-supine position) within normal range of the clinical site, or outside the normal range and not considered clinically significant by the Investigator.
   * Standard 12-lead ECG parameters (recorded after resting for 5 minutes in semi-supine position) in the following ranges; QTc (Fridericia algorithm recommended) ≤ 450 ms for males and 470 ms for females, and normal ECG tracing, or abnormal ECG tracing not considered clinically relevant by the Investigator.
   * Laboratory parameters demonstrating no clinically significant abnormalities, as determined by the Investigator. Total bilirubin outside the normal range may be acceptable if total bilirubin does not exceed 1.5x ULN with normal conjugated bilirubin (with the exception of a patient with documented Gilbert syndrome).
4. A negative result on a urine drug screen and a repeat negative result on Day -1 (amphetamines/methamphetamines, barbiturates, benzodiazepines, cannabinoids, cocaine, opiates).
5. Female participants must not be pregnant or breastfeeding and must use an effective contraception method (as described in Section 4.4.3), with the exception of participants who have undergone sterilization more than 3 months prior to screening, or who are postmenopausal.

   A woman of childbearing potential (WOCBP) must undergo pregnancy testing prior to the first dose of the study drug. The participant must be excluded from the study if the serum pregnancy test is positive.

   A postmenopausal state is defined as 12 months of amenorrhea without an alternative medical cause. In the absence of 12 months of amenorrhea, menopause may be confirmed by Follicle-Stimulating Hormone (FSH) measurement (> 40 IU/L or mIU/mL).

   Females on HRT (Hormonal Replacement therapy), where menopausal status is indeterminate, will be required to use a non-estrogen hormonal contraceptive method if they wish to continue their HRT during the study. Participants must otherwise discontinue HRT to allow for confirmation of postmenopausal status prior to enrollment in the study.

   Regulation
6. Provide written informed consent prior to undertaking any study-related procedures.
7. Must not be under any administrative or legal supervision or under institutionalization as per a regulatory or juridical order.

Exclusion Criteria:

Participants who meet any of the following criteria will be excluded from the study:

Medical history and clinical status

1. Any history or presence of clinically relevant cardiovascular, pulmonary, gastrointestinal, hepatic, renal, metabolic, hematological, neurological, musculoskeletal, rheumatological, psychiatric, systemic, ocular, or infectious disease, or signs of acute illness.
2. Frequent severe headaches and/or migraines, recurrent nausea and/or vomiting (defined as vomiting more than twice a month).
3. Made a blood or plasma donation of ≥500 ml within 1 month prior to the first dose.
4. Demonstrated clinically significant (required intervention, e.g., emergency room visit, epinephrine administration) allergic reactions, which in the opinion of the Investigator, would interfere with the volunteer's ability to participate in the trial.
5. Known hypersensitivity to any component of the IMP formulation.
6. History or presence of drug or alcohol abuse (defined as alcohol consumption of more than 2 units per day on a regular basis).
7. Regular smoking (defined as more than 5 cigarettes or equivalent per week), or unable to stop smoking during the study. Occasional smokers may be enrolled but need to abstain during admission to the site.
8. Excessive consumption of beverages containing xanthine bases (defined as more than 4 glasses per day).

   Interfering substances
9. Any medication, including St John's Wort, within 14 days prior to administration of the first dose or within 5 times the elimination half-life or pharmacodynamic half-life of the medication, with the exception of hormonal contraception, menopausal hormone replacement therapy, or occasional paracetamol at doses up to 2 g/day.
10. Any consumption of grapefruit or products containing grapefruit within 5 days prior to the first dose administration.
11. Any vaccination in the 2 weeks prior to administration of the first dose (Covid19 vaccination included, and planned COVID19 vaccinations, including booster shots, during the study or for 2 weeks after the last dose of study drug).

    General conditions
12. Any participant who, in the judgment of the Investigator, is likely to be non-compliant during the study, or to be unable to cooperate due to language problems or poor mental development.
13. Any participant who enrolled in or participated in any other clinical study involving an investigational medicinal product, or in any other type of medical research within 1 month or within 5 times the elimination half-life prior to administration of the first dose.
14. Any participant who cannot be contacted in the case of an emergency.
15. Any participant who is the Investigator or any subinvestigator, research assistant, pharmacist, study coordinator, or other staff thereof directly involved in conducting the study or any person dependent on (employees or immediate family members) the study site, the Investigator or the Sponsor.

    Biological status
16. Positive result on any of the following tests: hepatitis B surface antigen (HBsAg), hepatitis B core antibodies (HBcAb), anti-hepatitis C virus antibodies (anti-HCV), anti-human immunodeficiency virus 1 and 2 antibodies (anti-HIV1 and anti-HIV2 Ab).
17. Positive alcohol test at D-1.
18. Any participant in whom venous blood collection is difficult.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 66 (Estimated)
Dates: Start 2024-02-24 (Actual); Primary Completion 2025-02-28 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Part A-Single ascending dose: Incidence of AE, especially greater than Grade 2(CTCAE 5.0) | Up to 8 days
  Safety: Incidence of AE, especially greater than Grade 2(CTCAE 5.0)
Part B-multiple ascending dose (MAD): Incidence of AE, especially greater than Grade 2(CTCAE 5.0) | Up to 17 days
  Safety: Incidence of AE, especially greater than Grade 2(CTCAE 5.0)
Part A-Single ascending dose: Incidence of termination of taking IP | Up to 6-8 days
  Tolerability:Incidence of termination of taking IP
Part B-multiple ascending dose: Incidence of termination of taking IP | Up to 17 days
  Tolerability:Incidence of termination of taking IP

SECONDARY OUTCOMES:
Part A-Single ascending dose (SAD):Maximum Plasma Concentration (Cmax) | Up to 6-8 days
  PK parameters:Maximum Plasma Concentration [Cmax]
Part A-Single ascending dose (SAD): Area under the plasma concentration versus time curve (AUC) | Up to 8 days
  PK parameters (under food effect): Area Under The Curve (AUC)
Part A-Single ascending dose (under food effect):Maximum Plasma Concentration (Cmax) | Up to 8 days
  PK parameters (under food effect): Peak Plasma Concentration (Cmax)
Part A-Single ascending dose (under food effect): Area under the plasma concentration versus time curve (AUC) | Up to 8 days
  PK parameters (under food effect): Area under the plasma concentration versus time curve (AUC)
Part B- Multiple ascending dose (MAD):: Maximum Plasma Concentration [Cmax | Up to 17 days
  To assess the PK parameters of IPG11406 after ascending multiple oral doses

CONTACTS AND LOCATIONS:
Locations (1):
- Zhejiang Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No